CLINICAL TRIAL: NCT02205346
Title: Urinary Leukotriene E4 Levels in Children With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Medarva (Unknown)
Responsible Party: Sponsor
Other Study IDs: October 2013
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment

SUMMARY:
Investigate urinary leukotriene E4 levels and determine if there is a correlation with severity of obstructive sleep apnea. The investigators then would like to determine a threshold level which could then be used for confirmation of diagnosis of obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* children 2-16 years of age
* scheduled for polysomnogram

Exclusion Criteria:

* cardiovascular, neuromuscular, immunologic or craniofacial disorders
* pharmacologic treatment including corticosteroids and leukotriene receptor antagonists in the last month
* subjects who have already received treatment for OSA with an oral appliance, continuous positive airway pressure (CPAP) device
* previously undergone tonsillectomy and/or adenoidectomy

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Otolaryngology practice
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
urine leukotriene level | baseline
  assess urinary leukotriene E4 levels in children with obstructive sleep apnea (OSA

SECONDARY OUTCOMES:
correlation between Urine LTE4 and the apnea hypopnea index (AHI) | baseline
  determine if there is a correlation between urine LTE4 levels and the severity score as determined by the AHI

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Baldassari, MD, Principal Investigator — EVMS
Locations (1):
- Children's Hospital of the King's Daughters, Norfolk, Virginia, United States